CLINICAL TRIAL: NCT03747770
Title: A Community Intervention Effectiveness Study: Single Dose or Two Doses of Bivalent HPV Vaccine (CERVARIX) in Female School Students in Thailand
Brief Title: Effectiveness of Single Dose or Two Doses of Bivalent HPV Vaccine in Thailand
Acronym: IVIHPV1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Vaccine Institute (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IVI HPV1
Record Dates: First submitted 2018-11-11; First posted 2018-11-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: CERVARIX; Urine; DNA PCR; HPV infection; HPV genotyping; Effectiveness
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Age range of subjects: 13 up to 18 years of age
  * Vaccination - grade 8: 13 to less than 15 years of age
  * Behavioral questionnaire: grade 8 (as above) and 15-18 years of age for baseline (unvaccinated) and Year 2 and Year 4 cross-sectional surveys post vaccination
  * Urine collection: 15-18 years of age for baseline (unvaccinated) and Year 2 and Year 4 cross-sectional surveys post vaccination
  * Blood collection: grade 8 (as above) and 15-18 years of age for Year 2 and Year 4 cross-sectional surveys post vaccination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cross-sectional baseline survey (No Intervention): This are will collect behavioral questionnaire and urine in Grade 10 high school and Year 1 vocational school and Grade 12 high school and Year 3 Vocational school female students
- Single Dose HPV vaccination (Active Comparator): Grade 8 female students from Udon Thani Province This arm will collect behavioral questionnaire and blood prior vaccination Intervention: Single Dose HPV Vaccination with CERVARIX®(Glaxo Smith Kline, GSK, Rixensart, Belgium)
  Interventions: Biological: Bivalent HPV vaccine CERVARIX®
- Two-dose HPV vaccination (Active Comparator): Grade 8 female students from Buriram Province This arm will collect behavioral questionnaire and blood prior vaccination Intervention: Two-Dose HPV Vaccination with CERVARIX®(Glaxo Smith Kline, GSK, Rixensart, Belgium)
  Interventions: Biological: Bivalent HPV vaccine CERVARIX®
- Cross-sectional survey at Year 2 (No Intervention): This arm will collect behavioral questionnaire, urine and blood in Grade 10 high school and Year 1 vocational school female students
- Cross-sectional survey at Year 4 (No Intervention): Cross-sectional survey at Year 4 post vaccination

INTERVENTIONS:
Biological: Bivalent HPV vaccine CERVARIX® — Bivalent HPV vaccine(Glaxo Smith Kline, GSK, Rixensart, Belgium) presented as a suspension for intramuscular injection containing purified viral L1 protein for HPV types 16 and 18. Each 0.5 mL dose of the bivalent vaccine contains 20μg of HPV-16 L1 protein and 20 μg of HPV-18 L1 protein adsorbed onto a proprietary adjuvant system containing 500 μg of aluminum hydroxide and 50 μg of 3-O-desacyl-4-monophosphoryl lipid A (AS04)
  Arms: Single Dose HPV vaccination; Two-dose HPV vaccination

SUMMARY:
This is a community intervention effectiveness study in female school students in Thailand.

The study objectives are:

1. To demonstrate HPV vaccine effectiveness of Single Dose (SD) by a reduction in vaccine-type HPV prevalence (HPV 16 and HPV 18) at Year 2 and Year 4 post vaccination compared to unvaccinated same grade female students
2. To demonstrate that HPV vaccine effectiveness of SD and two-dose (2D) regimens are similar by comparing reductions in vaccine type prevalence at Year 2 and Year 4 post vaccination compared with the baseline surveys in the two provinces

DETAILED DESCRIPTION:
The study will investigate the effectiveness of a SD of HPV vaccine through the conduct of a regional effectiveness study in Thailand.

The study will be conducted in schools and district hospitals from the two selected provinces (Udon Thani and Buriram)

The study design includes 4 distinct and independent components:

1) vaccination, 2)baseline cross-sectional survey, 3,4)sequential cross-sectional surveys for impact assessments at Year 2 and Year 4 post vaccination.

* Vaccination: The target population is represented by all Grade 8 female students in the two provinces. All enrolled students will receive either SD (Udon Thani) or 2D (Buriram). A subset (N=200/province) of Grade 8 female students in each province will be selected for a blood collection before vaccination for assessment of vaccine immunogenicity.
* Surveys (baseline, Year 2 and Year 4 impact surveys): Target populations of are a subset of female students of Grades 10 High school (HS)/year 1 Vocational School (VS) and Grade 12 HS/year 3 VS from all schools in the two provinces and the sampling unit is an individual. Urine collection will be performed to assess HPV infection by DNA PCR and for genotyping of positive samples. A subset of students (N=200 per province) will be randomly selected for each of the Year 2 and Year 4 surveys for blood collection for assessment of vaccine immunogenicity.
* Demographics and sexual behavior questionnaire will be collected from all students.

ELIGIBILITY:
Inclusion criteria

A. Grade 8 (Mathayom 2):

1. Female students with identification card
2. Less than 15 years of age
3. Parent or guardian consent for vaccination and blood collection as applicable Participant assent for vaccination, questionnaire, and blood collection as applicable

B. Baseline survey (Grade 10 / year 1, Grade 12 / year 3)

1. Female students with identification card Participant assent for questionnaire and urine collection

C. Year 2 post vaccination survey( Grade 10 / year 1) Year 4 post vaccination survey (Grade 12 / year 3)

1. Female students with identification card
2. Parent or guardian consent for blood collection as applicable
3. Participant assent for questionnaire, urine and blood collection from those vaccinated at Grade 8 as applicable

Exclusion criteria

A. Grade 8 (Mathayom 2):

1. Students who already received HPV vaccination
2. Reported pregnancy
3. Any student who has a preexisting known medical condition or diagnosed psychological illness which in the opinion of the Principal Investigator or designee may be detrimental to her wellbeing

B. Baseline survey (Grade 10 / year 1, Grade 12 / year 3) 1. Any student who has a preexisting known medical condition or diagnosed psychological illness which in the opinion of the Principal Investigator or designee may be detrimental to her wellbeing

C. Year 2 post vaccination survey( Grade 10 / year 1) Year 4 post vaccination survey (Grade 12 / year 3)

1. Any student who has a preexisting known medical condition or diagnosed psychological illness which in the opinion of the Principal Investigator or designee may be detrimental to her wellbeing

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female students
Enrollment: 18000 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
HPV infection prevalence | Baseline survey (unvaccinated students) during the first year of the study
  HPV DNA PCR in urine
HPV infection prevalence | Year 2, two years post vaccination
  HPV DNA PCR in urine
HPV infection prevalence | Year 4, four years post vaccination
  HPV DNA PCR in urine
Identification of HPV circulating strains | Baseline survey (unvaccinated students) during the first year of the study
  HPV genotyping on urine positive samples
Identification of HPV circulating strains | Year 2, two years post vaccination
  HPV genotyping on urine positive samples
Identification of HPV circulating strains | Year 4, four years post vaccination
  HPV genotyping on urine positive samples

SECONDARY OUTCOMES:
HPV type-specific antibody response prior and post vaccination | Prior vaccination and at Year 2 and Year 4 Post vaccination
  Blood Sample

CONTACTS AND LOCATIONS:
Overall Officials: Suchada Jiamsiri, MD, Principal Investigator — Department of Disease Control, Thailand Ministry of Public Health, Bangkok
Locations (1):
- Ministry of Public Health, Bangkok, Chang Wat Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: No